CLINICAL TRIAL: NCT03841968
Title: Randomized Trial of Ultrasound-guided Right Internal Jugular Vein Catheterization Using Dynamic Short Axis Versus Conventional Long-axis View in Cardiac Surgery Patients: a Dual-center Randomized Trial
Brief Title: Dynamic SAX vs Conventional LAX in Internal Jugular Vein Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DNTP IJV
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Surgical Procedures; Central Venous Catheterization; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic needle tip positioning (Active Comparator): Dynamic needle tip positioning
  Interventions: Procedure: Dynamic needle tip positioning under ultrasound-guidance
- Conventional long-axis (Active Comparator): Conventional long-axis
  Interventions: Procedure: Conventional long-axis view

INTERVENTIONS:
Procedure: Dynamic needle tip positioning under ultrasound-guidance — The tip of needle is positioned under ultrasound-guidance using dynamic short-axis view.
  Arms: Dynamic needle tip positioning
Procedure: Conventional long-axis view — The tip of needle is positioned under ultrasound-guidance using conventional long-axis in-plane view.
  Arms: Conventional long-axis

SUMMARY:
Conventionally, short-axis out-of-plane (SAX) or long-axis in-plane (LAX) ultrasound views are commonly used to guide internal jugular vein catheterization.

SAX dynamic needle tip positioning (SAX-DNTP) is a novel ultrasound imaging technique that enables continuous visualization of the needle tip during ultrasound-guided cannulation; When the needle tip is imaged as a hyperechoic dot, the ultrasound probe is moved a few millimeters, and then the needle is advanced until the needle tip reappears in the vessel lumen. The process is repeated until the needle is advanced more than 1 cm into the lumen. The catheter is then introduced into the vessel.

The aim of this study was to compare the first pass success rate of internal jugular vein catheterization between SAX-DNTP and the conventional LAX technique.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery where central venous catheterization is required.

Exclusion Criteria:

* skin infection or trauma
* Shock
* Patients on ECMO or IABP support
* Morbid obesity
* Profound coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
First pass success rate of the internal jugular vein catheterization_confirmation of the central venous pressure through a patient monitor | Intraoperative
  First pass success rate of the internal jugular vein catheterization_confirmation of the central venous pressure through a patient monitor

SECONDARY OUTCOMES:
Total procedure time | Intraoperative
  Total procedure time
Rate of posterior wall puncture_assessed by ultrasound | Intraoperative
  Rate of posterior wall puncture_assessed by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea